CLINICAL TRIAL: NCT06463821
Title: Symptom Spectrum and Risk Factors for Fever in Pediatric and Adult Patients With Omicron Infection: a Prospective Observational Study
Brief Title: Symptom Spectrum and Risk Factors for Fever in Pediatric and Adult Patients With Omicron Infection
Status: Completed | Type: Observational
Sponsor: Shanghai Children's Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: SCMCIRB-K2022040-1
Record Dates: First submitted 2024-06-11; First posted 2024-06-18 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Symptom Spectrum and Risk Factors for Fever
Keywords: COVID-19, omicron, symptom spectrum, fever, vaccination, antipyretic
MeSH Terms: conditions — COVID-19; Fever

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- pediatric patients: pediatric patients who attended the child-parent sections of the Fangcang shelter hospitals with laboratory-confirmed COVID-19
  Interventions: Other: observational questionnaires
- adult patients: adult patients who attended the child-parent sections of the Fangcang shelter hospitals with laboratory-confirmed COVID-19
  Interventions: Other: observational questionnaires

INTERVENTIONS:
Other: observational questionnaires — Patient data were collected from questionnaires.

SUMMARY:
The omicron variant of coronavirus disease 2019 (COVID-19) has caused a global epidemic in 2022. The aim was to investigate the symptom spectrum and risk factors for fever in pediatric and adult patients with omicron infection. From April 8, 2022 to May 17, 2022, this prospective observational study included patients who attended the child-parent sections of the Fangcang shelter hospitals with laboratory-confirmed COVID-19. Patient data were collected from questionnaires. The risk factors for prolonged fever and high fever were identified by univariate and multivariate analyses.

DETAILED DESCRIPTION:
Study design and participants A prospective multicenter study was designed. It was conducted in accordance with the Declaration of Helsinki (as revised in 2013). Informed consent was obtained for all participants. From April 8, 2022 to May 17, 2022, Patients who attended the child-parent sections of the Fangcang shelter hospitals in Shanghai, China, with laboratory-confirmed COVID-19 were included. Those who had poor compliance (defined as inability to comply with the protocol) were excluded. Data from the included cases were collected. Adult patients and caregivers of children patients received two kinds of questionnaires after admission. Type I questionnaire (supplemental material) for basic characteristic were finished as soon as they were admitted. Type II questionnaire (supplemental material) for symptom and medication use tracking were filled out every day until discharge. This study was approved by the ethics committee of Shanghai Children's Medical Center.

Definition of outcomes The outcomes were the likelihood of developing prolonged fever and the likelihood of developing high fever. Fever was defined as temperature ≥ 38.0℃. Prolonged fever was defined as fever for more than 2 days. High fever was defined as temperature ≥ 39.1℃.

Statistical analysis SPSS version 25.0 (IBM SPSS Statistics, Armonk, NY, USA) was used to analyze the data. Data are presented as median values and interquartile ranges (IQRs) for continuous variables and frequencies and percentages for categorical variables. The investigators used Mann-Whitney U test to compare continuous variables between two groups. The investigators used χ2 test or Fisher exact test to compare categorical variables. Univariable analysis was used to investigate the association of each clinical variable with the outcomes. To determine the risk factors for each outcome, multivariable analysis was performed by logistic regression with a stepwise variable model. Variables of P value < 0.05 were candidates for multivariable analysis. Statistical significance was determined as a 2-sided P value of < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* hospitalized in the child-parent sections of the Fangcang shelter hospitals in Shanghai, China
* diagnosis of laboratory-confirmed COVID-19

Exclusion Criteria:

● have poor compliance (defined as inability to comply with the protocol)

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who attended the child-parent sections of the Fangcang shelter hospitals in Shanghai, China, with laboratory-confirmed COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 2591 (Actual)
Dates: Start 2022-04-08 (Actual); Primary Completion 2022-05-17 (Actual); Study Completion 2022-05-17 (Actual)

PRIMARY OUTCOMES:
Number of Participants with prolonged fever or high fever | From April 8, 2022 to May 17, 2022
  Fever's defined as temperature ≥ 38.0℃. Prolonged fever's defined as fever for more than 2 days. High fever's defined as temperature ≥ 39.1℃. Questionnaires for basic characteristic're finished as soon as they're admitted. Questionnaires for symptom and medication use tracking're filled out every day until discharge. The risk factors for prolonged fever and high fever're identified by univariate and multivariate analyses.

CONTACTS AND LOCATIONS:
Locations (1):
- child-parent sections of the Fangcang shelter hospitals, Shanghai, China

IPD SHARING:
Plan to Share IPD: No